CLINICAL TRIAL: NCT04274322
Title: Identifying Critically-ill Patients With COVID-19 Who Will Benefit Most From Nutrition Support Therapy: Validation of the NUTRIC Nutritional Risk Assessment Tool (COV_NUTRIC)
Brief Title: Identifying Critically-ill Patients With COVID-19 Who Will Benefit Most From Nutrition Support Therapy: Validation of the NUTRIC Nutritional Risk Assessment Tool
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: School of Pharmaceutical Sciences, Peking University, Beijing, China (Unknown); Department of Medicine, Queen's University, Kingston, Ontario, Canada (Unknown)
Responsible Party: Principal Investigator, Qinggang GE, M.D. Chief physician, Peking University Third Hospital
Other Study IDs: COV_NUTRIC
Record Dates: First submitted 2020-02-16; First posted 2020-02-18 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Critically Ill; Coronavirus Infections
Keywords: Critically Ill; Coronavirus Infections; Nutritional Risk; Nutrition; Intensive Care Unit
MeSH Terms: conditions — Critical Illness; Coronavirus Infections | interventions — Nutrition Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: High NUTRIC score
  Interventions: Other: Nutrition support
- Cohort 2: low NUTRIC score
  Interventions: Other: Nutrition support

INTERVENTIONS:
Other: Nutrition support — Calories and proteins are given to patients by using ways as parenteral nutriton, enteral nutrition, oral nutrition supplement

SUMMARY:
There was an interaction between mortality, nutritional intake and the Nutrition Risk in Critically ill (NUTRIC) score suggesting that those with higher NUTRIC scores benefited the most from increasing nutritional intake. Yet limited data were in Chinese patients. The current outbreak of novel coronavirus, named COVID-19, was first reported from Wuhan, China on Dec ember 31 , 2019. There are about 16% patients need ICU admission. The objective of this study is to validation of the "NUTRIC" nutritional risk assessment tool in Chinese ICU patients diagnosed as COVID-19.

DETAILED DESCRIPTION:
Heyland et al. previously proposed a novel scoring tool, the Nutrition Risk in Critically ill (NUTRIC) score, which is the first nutritional risk assessment tool developed and validated specifically for intensive care unit (ICU) patients. Many other risk scores and assessment tools exist to quantify nutrition risk but none have been specifically designed for ICU patients. Indeed, they generally consider all critically ill patients to be at high nutritional risk. However, the recognition that not all ICU patients will respond the same to nutritional interventions was the critical concept behind the NUTRIC score. There was an interaction between mortality, nutritional intake and NUTRIC score suggesting that those with higher NUTRIC scores benefited the most from increasing nutritional intake. However, the inferences about the validity of the NUTRIC score are limited in Chinese patients because of no data.

The current outbreak of novel coronavirus was first reported from Wuhan, China on Dec ember 31 , 2019 . This virus was named as 2019 nCoV by World Health Organization ( on Jan uary 12 , 2020). Following the advice of the Emergency Committee, the WHO declared the outbreak of 2019 nCoV a Public Health Emergency of International Concern . Patients show fever and / or respiratory symptoms, with the imaging characteristics of pneumonia, and other symptoms include hemoptysis muscle pain, headache, confusion, chest pain, and diarrhea. About 16% patients need ICU admission.

The objective of this study is to validation of the "NUTRIC" nutritional risk assessment tool in Chinese ICU patients diagnosed as COVID-19. This is a single-center, prospective cohort study of ICU patients with COVID-19. Data for all variables of the NUTRIC score will be collected. These include age, APACHE II score, SOFA score, number of co-morbidities, days from hospital admission to ICU admission. A logistic model including the NUTRIC score, the nutritional adequacy and their interaction will be estimated to assess if the NUTRIC score modified the association between nutritional adequacy and 28-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to intensive care unit (ICU), Peking University Third Hospital since Feb 2020
* Adult (aged over 18 years)
* Anticipate a length of ICU stay (LOS) of more than 48 hours
* Diagnosed as 2019 coronavirus disease (COVID-19)
* With food intake difficulties (can't intake food by oneself)

Exclusion Criteria:

* aged under 18 years
* Actual ICU LOS of less than 48 hours
* Using medications of IL-6 or IL-6R
* Overdose
* Written informed consent not obtained in the prospective cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The adult patients with 2019 coronavirus disease (COVID-19) admitted to ICU, Peking University Third Hopital from Feb 2020 to May 2020 will be involved in this study
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-04-04 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
28-day all cause mortality | from admission to 28-day/discharge, an average of length of ICU stay is 28-day

SECONDARY OUTCOMES:
All cause infection | from admission to 28-day/discharge, an average of length of ICU stay is 28-day
The rate of complications | from admission to 28-day/discharge, an average of length of ICU stay is 28-day
Length of ICU stay | from admission to 28-day/discharge, an average of length of ICU stay is 28-day
Duration of mechanical ventilation | from admission to 28-day/discharge, an average of length of ICU stay is 28-day

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No